CLINICAL TRIAL: NCT06214728
Title: Assesment of Changes ın Clinical and Radiographic Parameters Following the Application of Local Hyaluronic acıd Gel as an Adjunct to Minimally Invasive Non-surgical Treatment of Intraosseous Defects
Brief Title: Use of Hyaluronic Acid Gel in Intraosseous Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UGUNDOGDU1
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Periodontitis
Keywords: minimally invasive; nonsurgical periodontal debridements; periodontitis; alveolar bone loss; hyaluronic acid
MeSH Terms: conditions — Periodontitis; Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Subjects having more than one intrabony defect that meets the inclusion criteria, only one intraosseous defect per patient was included based on a preliminary randomisation by a coin toss (UGE). Patients were then block randomised and the allocation sequence was computer-generated using www.randomizer.org. The patient groups were recorded by another investigator who did not perform the treatment application and clinical measurements (SG).
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINST (Placebo Comparator): Minimally invasive non-surgical treatment (MINST): Using mini five curettes and ultrasonic devices with precise tips , the root surfaces were cleaned reaching to the base of the pocket, avoiding excessive root surface smoothing and gingival curettage.
  Interventions: Procedure: Placebo gel application
- MINST+HA (Active Comparator): Minimally invasive non-surgical technique (MINST) with application of Hyaluronıc Acid gel: Using mini five curettes and ultrasonic devices with precise tips , the root surfaces were cleaned reaching to the base of the pocket, avoiding excessive root surface smoothing and gingival curettage. HA gel was applied to the periodontal pockets where the intraosseous defect was located using a sterile injector with a plastic needle. The gel was applied until it overflowed from the gingival sulcus.
  Interventions: Procedure: Hyaluronic acid gel application

INTERVENTIONS:
Procedure: Hyaluronic acid gel application — HA gel was applied to the periodontal pockets where the intraosseous defect was located using a sterile injector with a plastic needle. The gel was applied until it overflowed from the gingival sulcus. Patients were instructed not to eat, drink or brush their teeth for at least one hour. Subgingival application of HA was repeated 4 weeks after the first session.
  Arms: MINST+HA
Procedure: Placebo gel application — The control group received placebo HA gel probe without rinsing. Placebo application was repeated 4 weeks after the first session.
  Arms: MINST

SUMMARY:
Aim:

The aim of this randomised, parallel-arm, blinded, controlled clinical trial was to compare the clinical and radiographic efficacy of MINST with and without 0.8% HA gel application in the treatment of intraosseous defects.

Research Hypothesis:

The null hypothesis that there is no statistically significant difference in clinical and radiographic measurements between the use of HA gel in addition to MINST for the treatment of intraosseous defects and MINST treatment alone was tested.

DETAILED DESCRIPTION:
This study was designed as a randomised controlled clinical trial and conducted between March 2022 and May 2023 at the Department of Periodontology, Bezmialem Vakıf University. Ethical approval was obtained from Clinical Research Ethics Committee of Bezmialem Vakıf University with approval number E.54753 on March 15, 2022.

The patients included in our study were selected from a total of 140 patients with complaints of gingival problems who applied to the Department of Periodontology at Bezmialem Vakıf University Faculty of Dentistry, specifically those having intraosseous defects in the premolar/molar teeth. Forty-two individuals were included in the study, and it was completed with a total of 36 participants, consisting of 25 females and 11 males.

Initial clinical periodontal measurements and periapical radiographs were taken from the defect area with parallel technique in the first session. Occlusal stents with fixed guide points were prepared to place the periodontal probe with the correct angle and inclination. During the initial session, complete oral supragingival calculus cleaning and oral hygiene motivation were performed. After that, patients were randomly assigned to the test (MINST + HA, n = 17) or control (MINST, n = 19) groups. Neither the patients nor the expert responsible for the clinical measurements (UGE) was aware of which treatment each individual had received.

The MINST concepts described by Nibali et al. were followed in the treatment protocol. During the procedure, a subpapillary approach was taken to reduce trauma to the soft tissues, particularly the papillae, using a 2.5x420 mm magnification loop . The instruments were gently placed within the periodontal pocket while the patient was under local anaesthesia , in order to keep the soft tissues stable. Using mini five curettes and ultrasonic devices with precise tips ,the root surfaces were cleaned reaching to the base of the pocket, avoiding excessive root surface smoothing and gingival curettage. The subgingival area was not irrigated to prevent deterioration of clot stabilisation during the wound healing process [1]. MINST was performed in all areas of the oral cavity with periodontal pockets >3 mm. The control group was treated with MINST alone without using any irrigation solution. Beside, in the test group, following MINST protocol same as in the control, HA gel was applied to the periodontal pockets where the intraosseous defect was located using a sterile injector with a plastic needle. The gel was applied until it overflowed from the gingival sulcus. Patients were instructed not to eat, drink or brush their teeth for at least one hour. Subgingival application of HA was repeated 4 weeks after the first session. The control group received placebo HA gel probe without rinsing.

Clinical examination Initial clinical measurements were taken by a single investigator (UGE) using the UNC15 probe at six sites on all teeth to determine the stage and grade of periodontitis in study population.

Clinical periodontal measurements of the defect site were recorded at baseline and repeated at 3 and 6 months following treatment. Probing depth (PD), clinical attachment level (CAL) and gingival recession (GR) measurements were made from two points including buccal and lingual area through a patient-specific acrylic stent in the defect area and recorded as average and deepest/worst. Bleeding on probing (BoP) and presence of plaque (P) were evaluated as present/absent in the buccal and lingual part of the defect area and recorded as %.

The gingival phenotype was evaluated by observing the probe's silhouette visibility using biotype probe located in the buccal point of the intraosseous defect area.

Pre-study investigator calibration was performed by repeating the PD and CAL measurements of 10 periodontitis patients who were not included in the study at 24 hours intervals. The intraclass correlation showed that the researcher's repeatability was at an acceptable level (PD; k-score: 0,817-0,952; CAL:0,836-0,926).

Radiographic examination For the diagnosis of intraosseous defects radiographs were taken at baseline and 6-month follow-up using a custom-made radiographic stent and the parallel cone technique. Radiographs were digitized and analysed by a single calibrated investigator using a computer software (Planmeca Romexis Viewer software). The radiographs were numbered prior to analysis to blind the analyst to the groups of radiographs. For investigator calibration, measurements of intraosseous defect depth (infra) and defect angle of periapical radiographs from 10 nonstudy patients were repeated at 24-hour intervals. Intra-class correlation coefficients ranging from 0.86 to 0.92 for the defect depth and angle measurements and it was determined that the reproducibility of the researcher was at an acceptable level. Radiographic measurements were made by using the reference points on tooth surface. Total defect depth (TDD): The distance from the cemento- enamel junction to the base of the defect (CEJ-DD) was measured. Intraosseous defect depth (INFRA): It is the distance from the projection of the alveolar crest point on the tooth to the bottom of the defect (DD). Distance from the CEJ to the alveolar crest (CEJ-BC): It is the distance from the projection of the alveolar crest point on the tooth and the cemento enamel junction (CEJ). Intra-osseous defect angle: The radiographic defect angle was measured between the CEJ-BD line of the involved tooth and the bone defect surface.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe/progressed periodontitis (stage III/IV)
* Presence of an intraosseous defect with a probing depth ≥ 5 mm and defect depth ≥ 3 mm;
* Absence of furcation involvement,mobility and subgingival restoration in the vital tooth with intraosseous defect.

Exclusion Criteria:

* Systemic diseases
* Smokers
* Pregnant or lactating women
* Those who received periodontal treatment within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Intraosseous defect depth (INFRA) | Baseline - 6 months
  It is the distance from the projection of the alveolar crest point on the tooth to the bottom of the defect (DD)

SECONDARY OUTCOMES:
Probing depth (PD) | Baseline - 3months - 6 months
  as the measurement of the length between the bottom of the periodontal pocket to marginal gingiva
Clinical attachment level (CAL) | Baseline - 3months - 6 months
  distance between the base of the pocket and the enamel cement junction

OTHER OUTCOMES:
Gingival recession (GR) | Baseline - 3months - 6 months
  as the measurement of the distance between the marginal gingiva and cemento-enamel junction
Bleeding on probing (BoP) | Baseline - 3months - 6 months
  present/absent in the buccal and lingual part of the defect area and recorded as %.
Plaque (P) | Baseline - 3months - 6 months
  present/absent in the buccal and lingual part of the defect area and recorded as %.
Total defect depth (TDD) | Baseline - 6 months
  The distance from the cemento- enamel junction to the base of the defect (CEJ-DD) was measured.
Distance from the CEJ to the alveolar crest (CEJ-BC) | Baseline - 6 months
  It is the distance from the projection of the alveolar crest point on the tooth and the cemento enamel junction (CEJ).
Intra-osseous defect angle | Baseline - 6 months
  The radiographic defect angle was measured between the CEJ-BD line of the involved tooth and the bone defect surface

CONTACTS AND LOCATIONS:
Overall Officials: Sadiye Gunpinar, Asc. Prof., Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)